CLINICAL TRIAL: NCT00416663
Title: A Study for Testing Efficacy and Safety of the Administration of Vescell(TM) (Blood-Borne Autologous Angiogenic Cell Precursors) to Alleviate Anginal Symptoms and Myocardial Ischemia in Severe Anginal Syndrome +/- Heart Failure
Brief Title: Vescell(TM) for the Treatment of Patients With Severe Anginal Syndrome With or Without Heart Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TheraVitae Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV-013
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2006-12

CONDITIONS: Angina Pectoris
Keywords: Stem cells; Progenitor cells; Angina Pectoris; Heart Failure; Angiogenesis
MeSH Terms: conditions — Angina Pectoris; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): open label,single arm,intervention is Angiogenic Cell Precusors(ACPs)
  Interventions: Procedure: Intracoronary administration of autologous ACPs

INTERVENTIONS:
Procedure: Intracoronary administration of autologous ACPs — Stem cells type:ACPs. At least 1.5 million of ACPs per one time of treatment
  Other Names: VescellTM

SUMMARY:
Evaluation of an intracoronary injection of ex-vivo generated autologous Angiogenic Cells Precursors (ACPs) to treat patients suffering from severe angina not responsive to maximal drug treatment or not willing or without option of undergoing percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG). The use of ACPs aims to promote the formation of new vascularization and thus viable myocardial tissue.

DETAILED DESCRIPTION:
Ten adult patients with severe angina pectoris with or without heart failure and no therapeutic alternative will undergo screening and be treated with an injection of Angiogenic Cell Precursors (ACPs), contained in VesCell (TM). 250 ml of blood will be drawn from the patient and from this blood sample progenitor cells will be generated and differentiated into ACPs. The product will be administered into the obstructed coronary arteries using a catheter. Following injection, patients will be hospitalized for 24-48 hours in intensive care and later as required by their medical condition. Patients will return for follow up testing at one, three and six months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic stable angina on maximal medical therapy and an occluded coronary artery or bridging collaterals to a patent distal segment supplying an ischemic viable myocardial region as shown on Sestamibi scan. On coronary angiography, the occluded coronary artery or bridging collaterals must have a patent proximal segment of at least 30 mm with at least one side branch to enable the injection of the VesCellTM if the vessel remains occluded despite the attempted angioplasty efforts (prior to or during the study angiography).
* Patients with occluded target coronary artery (with or without bridging collaterals) that could not be treated with PCI.
* Patients are not candidates for or are not willing to undergo CABG surgery.
* Age 18 to 80 years
* Male or non-pregnant, non-lactating female
* Ejection fraction >35% on Sestamibi
* Sestamibi scan (myocardial perfusion) during exercise or dipyridamole, demonstrating regional reversible ischemia in an area relating to the occluded coronary artery.
* Informed consent obtained and consent form signed

Exclusion Criteria:

* Patients not satisfying the coronary angiography and Sestamibi criteria.
* Patient who received blood transfusions during the previous 4 weeks (to exclude the potential of non-autologous ACPs in the harvested blood).
* Inability to communicate (that may interfere with the clinical evaluation of the patient)
* STEMI during the preceding 3 months
* PCI+stenting during the preceding three months
* Significant valvular disease or after valve replacement
* After heart transplantation
* Cardiomyopathy
* Renal failure (creatinine 10% above the upper limit according to the hospital normograms)
* Hepatic failure
* Anemia (lower than 11mg/dl.hemoglobin for female and lower than 12 mg/dl for male)
* Abnormal coagulation tests normal [platelets, PT (INR), PTT]
* Stroke within the preceding 3 years
* Malignancy within the preceding 3 years
* Concurrent chronic or acute infectious disease
* Severe concurrent medical disease (e.g., septicemia, HIV-1,2/HBV/HCV infections, insulin-dependent diabetes mellitus, systemic lupus erythematosus, multiple sclerosis, amyotrophic lateral sclerosis)
* Chronic immunomodulating or cytotoxic drugs treatment
* Patients who have rectal temperature above 38.40C for 2 consecutive days
* Patient unlikely to be available for follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-08; Study Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
Safety of the procedure as manifested in the post treatment observation and | 6 months
tests. | 6 months

SECONDARY OUTCOMES:
Changes from baseline to 1, 3 and 6 months in the CCS. | 6 months
Changes from baseline to 1, 3 and 6 months of modified Bruce exercise test. | 6 months
Changes from baseline to 6 months of exercise-induced ischemia on Sestamibi scan. | 6 months
Changes from baseline to 6 months of %LVEF | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan Tzivoni, MD, Principal Investigator — Director, Department of Cardiology, Shaare Zedek Medical Center, Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Porat Y, Porozov S, Belkin D, Shimoni D, Fisher Y, Belleli A, Czeiger D, Silverman WF, Belkin M, Battler A, Fulga V, Savion N. Isolation of an adult blood-derived progenitor cell population capable of differentiation into angiogenic, myocardial and neural lineages. Br J Haematol. 2006 Dec;135(5):703-14. doi: 10.1111/j.1365-2141.2006.06344.x. PMID 17052254